CLINICAL TRIAL: NCT02282748
Title: Swiss Longitudinal Cohort
Status: Recruiting | Type: Observational
Sponsor: Hypertension Excellence Centre Lucerne (Other)
Responsible Party: Sponsor
Other Study IDs: SNCTP 000000612
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
The planned research project is a prospective population-based cohort study, similar to the well-known Framingham study in the United States. So far, there is no similar research project in Switzerland.

It is planned to examine of three Swiss municipalities. Recruitment in a first Swiss municipality (Lostallo/Cama GR) started 2014 and ended in 2019. Overall, 496 participants were recruited in this municipality. The five-year follow-up in this municipality started in 2019. It is planned to start recruitment in a second Swiss municipality (Uznach SG) in 2020.

The examinations embrace a broad spectrum of measurements (for details the investigators refer to the published study protocol).

ELIGIBILITY:
Inclusion Criteria:

* Resident of Cama GR, Lostallo GR, or Uznach SG
* Age ≥6 years (no upper age limit), for voluntary blood sample ≥18 years
* Willing to participate in long-term study
* Written informed consent (in participants ≥6 years and <18 years signed by parents)

Exclusion Criteria:

* No exclusion criteria

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population of four Swiss municipalities
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-10; Primary Completion 2024-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 10 years

SECONDARY OUTCOMES:
Cardiovascular events | 10 years
  Cardiovascular events (i.e. stroke, myocardial infarction) will be assessed using questionnaires and case records.
Heart function | 10 years
  Heart function will be assessed using questionnaires for symptoms, clinical examination and measurement of electromechanical activation time.
Cognitive function | 10 years
  Cognitive function will be assessed using validated instruments.
Kidney function | 10 years
  Kidney function will be assessed using laboratory measurements.
Autonomy | 10 years
  Autonomy wil be assessed using validated instruments.
Nursing home admission | 10 years
  Nursing home admissions will be assessed using standardized questions.

OTHER OUTCOMES:
Changes in cardiovascular risk factors | 10 years
  Cardiovascular risk factors will be assessed using validated measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Study Chair — Hypertension Excellence Centre Lucerne; Andreas W Schoenenberger, MD, Principal Investigator — University Department of Geriatrics, University of Bern; Paolo Suter, MD, Principal Investigator — University of Zurich; Franco Muggli, MD, Principal Investigator — Swiss Society of Hypertension; Renate Schoenenberger, MD, Principal Investigator — Hypertension Excellence Centre Lucerne; Pierre-Alexandre Krayenbühl, MD, Principal Investigator — Linth Hospital
Locations (3):
- Switzerland (3):
  - Linth Hospital, Uznach, Canton of St. Gallen
  - Cama, Cama, Kanton Graubünden
  - Lostallo, Lostallo, Kanton Graubünden

REFERENCES:
- [Derived] Pusterla L, Radovanovic D, Muggli F, Erne P, Schoenenberger AW, Schoenenberger-Berzins R, Parati G, Suter P, Lava SAG, Gallino A, Bianchetti MG. Impact of Cardiovascular Risk Factors on Arterial Stiffness in a Countryside Area of Switzerland: Insights from the Swiss Longitudinal Cohort Study. Cardiol Ther. 2022 Dec;11(4):545-557. doi: 10.1007/s40119-022-00280-8. Epub 2022 Sep 24. PMID 36152116
- [Derived] Schoenenberger AW, Radovanovic D, Muggli F, Suter PM, Schoenenberger-Berzins R, Parati G, Bianchetti MG, Gallino A, Erne P. Prevalence of ideal cardiovascular health in a community-based population - results from the Swiss Longitudinal Cohort Study (SWICOS). Swiss Med Wkly. 2021 Sep 28;151:w30040. doi: 10.4414/smw.2021.w30040. eCollection 2021 Sep 27. PMID 34581550
- [Derived] Schoenenberger AW, Muggli F, Parati G, Gallino A, Ehret G, Suter PM, Schoenenberger-Berzins R, Resink TJ, Erne P. Protocol of the Swiss Longitudinal Cohort Study (SWICOS) in rural Switzerland. BMJ Open. 2016 Nov 28;6(11):e013280. doi: 10.1136/bmjopen-2016-013280. PMID 27895066